CLINICAL TRIAL: NCT07229638
Title: An Open-label, Multicenter Phase IB/II Clinical Study on the Safety, Tolerability, and Efficacy of SHR-9839(sc) in Combination Anti-tumor Therapy in Patients With Solid Tumors
Brief Title: A IB/II Phase Clinical Study on the Safety, Tolerability, and Efficacy of SHR-9839(sc) in Combination Anti-tumor Therapy in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-9839-202
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): SHR-9839(sc) combined with antitumor drugs.
  Interventions: Drug: SHR-9839(sc) For Injection

INTERVENTIONS:
Drug: SHR-9839(sc) For Injection — SHR-9839(sc) for injection.

SUMMARY:
This study is an open-label, multi-center Phase IB/II clinical trial of SHR-9839(sc) combined with anti-tumor therapy in patients with advanced solid tumors, aimed at evaluating the safety, tolerability, and efficacy of SHR-9839(sc) in combination with anti-tumor therapy in patients with advanced solid tumors. Phase IB is the dose escalation stage, and Phase II is the efficacy expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent, has signed the IRB/EC-approved informed consent form with the date indicated, and is willing and able to comply with treatment plan visits, examinations, and other procedural requirements;
2. Age 18-70 years (inclusive) at the time of signing the informed consent form, no gender restriction;
3. ECOG performance status of 0 or 1;
4. Expected survival ≥12 weeks;
5. At least one measurable lesion according to RECIST v1.1 criteria;
6. Subjects must provide at least 8 formalin-fixed, paraffin-embedded tumor tissue blocks or unstained tumor specimens. For subjects unable to provide tumor tissue as required, enrollment should be determined after discussion with the sponsor;
7. Major organ function must meet standards (no use of blood components or growth factors within 14 days before the first dose to correct abnormalities); test results must be completed within 7 days prior to the first study treatment;
8. Female subjects of reproductive potential must agree to use highly effective contraception starting from the signing of the informed consent form, throughout the study treatment period, and for 9 months after the last administration of the investigational product, and must avoid donating eggs during this period. Male subjects with partners of reproductive potential must agree to use highly effective contraception starting from the first dose of the investigational product, throughout the study treatment period, and for 6 months after the last administration of the investigational product, and must avoid donating sperm during this period. Female subjects must not be breastfeeding and must have a negative serum human chorionic gonadotropin (HCG) test within 7 days before the first dose (if the serum pregnancy test is positive, pregnancy must be excluded and enrollment confirmed after discussion with the sponsor).

Exclusion Criteria:

1. Patients with active central nervous system (CNS) metastases or leptomeningeal metastases (including a history of such);
2. Patients with other malignancies within 3 years before the first dose, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, locally resected prostate cancer, ductal carcinoma in situ post-surgery, or papillary thyroid carcinoma post-surgery (hormonal therapy for non-metastatic prostate or breast cancer is allowed);
3. Patients deemed by the investigator to have uncontrolled tumor-related pain. Subjects requiring analgesic treatment must have a stable analgesic regimen before entering the study; symptomatic lesions suitable for palliative radiotherapy should be treated prior to study entry;
4. Patients with severe cardiovascular or cerebrovascular disease;
5. Patients with clinically symptomatic moderate or severe ascites (i.e., requiring therapeutic paracentesis or drainage within 2 weeks before the study treatment; subjects with only minimal ascites shown on imaging without clinical symptoms may be enrolled); uncontrolled or moderate-to-large pleural effusion or pericardial effusion;
6. Patients with a history of interstitial pneumonia, including idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, radiation-induced pneumonia requiring steroid treatment, or those with suspected interstitial pneumonia on imaging at screening, or in whom interstitial pneumonia cannot be excluded (subjects with only fibrotic radiation pneumonitis in the radiation field may participate); or patients with respiratory failure, severe asthma, severe chronic obstructive pulmonary disease, or other serious lung diseases significantly affecting pulmonary function; or those who have previously undergone total lung resection;
7. Patients with severe infection within 4 weeks before the start of study treatment, including but not limited to bacteremia, severe pneumonia, or other serious infection complications requiring hospitalization; active infections of CTCAE grade ≥2 requiring systemic antibiotic therapy within 2 weeks before the first dose; subjects receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection) may be enrolled;
8. History of immunodeficiency, including positive HIV test; presence of active hepatitis B (HBsAg positive during the screening period, and DNA quantification ≥1000 copies/ml or 500 IU/ml) or hepatitis C (anti-HCV positive and HCV RNA positive);
9. Active pulmonary tuberculosis infection within one year prior to enrollment as indicated by medical history or imaging, or a history of active pulmonary tuberculosis more than one year ago that was not formally treated;
10. Previous adverse reactions to anti-tumor treatments that have not recovered to CTCAE ≤ grade 1 (except for alopecia, grade 2 peripheral neuropathy meeting the enrollment criteria, or other situations judged by the investigator not to affect study drug treatment);
11. Systemic anti-tumor treatment (including chemotherapy, biological therapy, targeted therapy, immunotherapy, radical radiotherapy, etc.) within four weeks prior to starting the study treatment;
12. Chest radiotherapy >30 Gy within 24 weeks prior to first use of the study drug, non-chest radiotherapy >30 Gy within four weeks prior to first use (subjects who completed brain metastasis radiotherapy within 14 days prior to first dose may be enrolled), and palliative radiotherapy ≤30 Gy within 14 days prior to first use;
13. Major organ surgery within 4 weeks prior to first use of the study drug (excluding biopsy), significant trauma, or planned elective surgery during the trial; minor traumatic surgery (biopsy, endoscopy, and drainage procedures) within seven days prior to first use of the study drug;
14. Within 3 months prior to the start of the study, participants who had intestinal obstruction or symptoms and signs of intestinal obstruction are excluded. However, if they have undergone surgical or other treatments and the obstruction has been completely relieved, they may be screened; those who have previously received intestinal stent placement and whose stent has not been removed by the screening period are also excluded;
15. Severe gastrointestinal disorders, including but not limited to grade ≥2 inflammation, diarrhea, bleeding, obstruction, perforation, or fistula (except for hemorrhoidal bleeding or cases presenting only as positive fecal occult blood, which may be included);
16. Use of live attenuated vaccines within 28 days before the first administration of the study drug, or anticipated need for live attenuated vaccines during the study treatment;
17. Pregnant or breastfeeding women, or women planning to become pregnant during the study period and within 7 months after the last administration of the study drug;
18. History of severe allergic reactions to any component of the proposed study drug;
19. According to the investigator's judgment, participants who have other factors that may affect the study results or potentially lead to premature termination of the study, such as alcoholism, drug abuse, other severe diseases (including psychiatric disorders) requiring concomitant treatment, severe laboratory abnormalities, domestic or social factors, and other circumstances that may impact participant safety or the collection of study data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | 28 days.
Adverse events (AEs) | 13 months.
Recommended Phase 2 Dose (RP2D) | From the first dose to the last visit, about 13 months.
Objective Response Rate (ORR) | From the first dose to the last visit, about 13 months.

SECONDARY OUTCOMES:
Disease control rate (DCR) | From the first dose to the last visit, about 13 months.
Duration of response (DoR) | From the first dose to the last visit, about 13 months.
Progression-Free Survival (PFS) | From the first dose to the last visit, about 13 months.
Overall Survival (OS) | From the first dose to the last visit, about 13 months.
Serious adverse events (SAEs) | From the first dose to the last visit, about 13 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Affiliated Cancer Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided